CLINICAL TRIAL: NCT03151538
Title: Assessment Effects on Pes Planus and Femoral Anteversion Angle of Exercise Training Mixed With Play on Pre-school Children
Brief Title: Effects on Pes Planus Exercise Training Mixed With Play on Pre-school Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burcu Talu (Other)
Responsible Party: Sponsor-Investigator, Burcu Talu, Assistant Professor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-54
Record Dates: First submitted 2017-04-26; First posted 2017-05-12 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Pes Planus; Flat Foot; Femoral Anteversion
Keywords: Pedography; Exercise; Play Training; Pes Planus; Femoral Anteversion
MeSH Terms: conditions — Flatfoot; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental, Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pes Planus Group (Experimental): This group of patients received children with pes planus. It will be applied exercise training mixed with play
  Interventions: Behavioral: Exercise Training Mixed With Play
- Controlled Group (Other): This group of patients received healthy children.
  Interventions: Other: Controlled

INTERVENTIONS:
Behavioral: Exercise Training Mixed With Play — To assess effects of training program which includes mixed exercises with playing.Study included 90 pre-school children who suffer from pes planus and increased femoral anteversion angle. Demographic data, navicular height, weight-bearing and non-weight bearing of subtalar joint motion, metatarsal width(weight and non-weight), range of hallux valgus,height of foot, tension of Achilles tendon, habits of W standing(hour/day), angle of Quadriceps(Q degree), angle of hip rotation were recorded . Craig Test, foot posture index, Chippaux-Smirak Index(CSI),Beighton hypermobility score, valgus index, thigh foot angle examination were used. CSI measurements were positive correlation with severity of pes planus.
  Arms: Pes Planus Group
Other: Controlled — First and last measurements will be done. There will be no intervention. Study will include 30 healthy pre-school children. Demographic data, navicular height, weight-bearing and non-weight bearing of subtalar joint motion, metatarsal width(weight and non-weight), range of hallux valgus,height of foot, tension of Achilles tendon, habits of W standing(hour/day), angle of Quadriceps(Q degree), angle of hip rotation were recorded . Craig Test, foot posture index, Chippaux-Smirak index(CSI),Beighton hypermobility score, valgus index, thigh foot angle examination were used.
  Arms: Controlled Group

SUMMARY:
The study was planned to assess effects on pes planus and femoral anteversion angle of exercise training mixed with play on pre-school children.

DETAILED DESCRIPTION:
Pes planus ( Pes planovalgus) is similar with flatfoot occurs collapse of medial longitudinal arch which is lower than normal range or occurs extra pressure on arch. It is separated two group such congenital (flexible and rigid) and acquired. The etiology of pes planus is that hallux rigidus, plantar calcaneonavicular ligament rupture, collapse of medial longitudinal arch, pathology of ligament and tendon, shortness Achilles tendon and juvenile hallux valgus. The most common causes of pes planus are outgroup of leg muscles (peroneal) spasticity, plantar fasciitis and tibial tendon insufficiency. Symptoms of pes planus are indicated heel pain, gait abnormalities, decreased dorsiflexion range of ankle, plantar ulceration, limited mobility of 1.metatarsophalangeal joint and spasm of peroneal muscle. There is a high prevalence rates among males and occur positive correlation between with pes planus and BMI. Evaluation methods of pes planus are X-ray, heel height, gait analysis and Achilles strain. The most commonly used method are line that medial malleolus, 1st metatarsal head and the navicula is on the same line, and the footprint technique from ink rubber plates. Treatment of pes planus is maintained medial displacement calcaneal osteotomy operation with the transfer of the flexor digitorum longus. Non- invasive treatment methods are given such as peroneal muscles and Achilles stretching exercises. 25 degree angle inverted foot orthoses are commonly used because of increasing stance phasic in treatment. Peroneal neural mobilization, play training and stretching exercises are often used treatment method of pes planus. Main purpose of this study is that assess effects of mixed training program with playing on pes planus and increased femoral anteversion angle in pre-school students.

ELIGIBILITY:
Inclusion Criteria:

* Children in an age range of 4-7 years,
* Having bilateral or unilateral deformity with pes planus
* CSI range > % 62.7 measured by the referring physical therapist.
* Having no any foot surgeon,
* Without any neurological diseases,
* Who want to be involved voluntary work,
* Pre-school students who have been informed by their families(their families approved illuminated affirmation ).

Exclusion Criteria:

* Pre-school students who can not adapt to training,
* Students who do not want to be involved in voluntary work.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Foot print with pedography (%). Change from pes planus at 6 week. | 6 weeks
  It used to define pes planus.

SECONDARY OUTCOMES:
Change from Angle of Quadriceps at 6 week. | 6 weeks
  The test used for angle of hip anteversion. (Degree)
Change from Valgus Index at 6 week. | 6 weeks
  It used to define pes planus. (Degree)
Change from Navicular Drop at 6 week. | 6 weeks
  It used to define pes planus. (mm)
Change from Angle of subtalar joint at 6 week. | 6 weeks
  It used to define pes planovalgus. (Degree)
Change from Craig test at 6 week. | 6 weeks
  The test used for angle of hip anteversion. (Degree)
Change from thigh foot angle examination at 6 week. | 6 weeks
  The test used for angle of tibial torsion. (Degree)

OTHER OUTCOMES:
Beighton Hypermobility Score | Baseline
  It used to define hypermobility.(Index score)

CONTACTS AND LOCATIONS:
Overall Officials: Burcu TALU, PhD, Principal Investigator — Inonu University
Locations (1):
- Preschool of Battalgazi and Yesilyurt district, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evans AM, Rome K, Carroll M, Hawke F. Foot orthoses for treating paediatric flat feet. Cochrane Database Syst Rev. 2022 Jan 26;1(1):CD006311. doi: 10.1002/14651858.CD006311.pub4. PMID 35080267
- [Derived] Evans AM, Rome K, Carroll M, Hawke F. Foot orthoses for treating paediatric flat feet. Cochrane Database Syst Rev. 2022 Jan 14;1(1):CD006311. doi: 10.1002/14651858.CD006311.pub3. PMID 35029841